CLINICAL TRIAL: NCT05809518
Title: Influence of Sedation Strategies on Hospital LOS and ICU LOS in Patients After Cardiac Surgery With Cardiac Pulmonary Bypass. Comparison of Propofol-based, Dexmedetomidine-based Sedation or Their Combination.
Brief Title: Influence of Sedation Strategies on Hospital LOS and ICU LOS in Patients Cardiac Surgery
Acronym: LOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anesthesia Research Group UA (Other)
Responsible Party: Principal Investigator, Plechysta Yelyzaveta, chief of the anesthesia department, Anesthesia Research Group UA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5-08-039.35
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Sedation Complication
Keywords: cardiac surgery; ICU sedation; hospital LOS; ICU LOS; vasopressors; postoperative sedation
MeSH Terms: interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Propofol Group (Experimental): Patient sedation after cardiac surgery at the intensive care unit.
  Sedation group (Pr):
  continuous infusion of propofol using a syringe pump at the dose of 1-1.5 mg / kg / h
  Interventions: Drug: Propofol injection
- Dexmedetomidine group (Experimental): Patient sedation after cardiac surgery at the intensive care unit.
  Sedation group Dexmedetomidine (Dx):
  continuous infusion of Dexmedetomidine using a syringe pump at the dose of 0.5-1.0 mcg/ kg / h
  Interventions: Drug: Dexmedetomidine injection
- Dexmedetomidine and propofol group (Experimental): Patient sedation after cardiac surgery at the intensive care unit.
  Sedation group DxPr:
  continuous infusion of propofol using a syringe pump at the dose of 0.5-1.5 mg / kg / h and dexmedetomidine 0.2-0.7 mcg\kg\h
  Interventions: Drug: Dexmedetomidine and Propofol

INTERVENTIONS:
Drug: Propofol injection — sedation after cardiac surgery
  Other Names: Pr
  Arms: Propofol Group
Drug: Dexmedetomidine injection — sedation after cardiac surgery
  Other Names: Dx
  Arms: Dexmedetomidine group
Drug: Dexmedetomidine and Propofol — sedation after cardiac surgery
  Other Names: DxPr
  Arms: Dexmedetomidine and propofol group

SUMMARY:
Preoperative, intraoperative and postoperative management of the patient are some of the main stages that can affect the hospital LOS and ICU LOS. Experience on the evidence-based approach and the progressive guidelines implementation of recommendations, the issue of the choice of drugs for sedation in the family and their impact on the length of stay in the intensive care unit and the length of hospitalization remain unsolved.

DETAILED DESCRIPTION:
Optimization of sedation regimes can become one of the factors that will help to reduce the length of hospital and ICU stay. The purpose of the study is to track is there a relationship between the drug for sedation and the length of stay of patients in the intensive care unit and in hospital treatment.

ELIGIBILITY:
Inclusion Criteria:

* Multi vascular lesions of the coronary arteries according to coronary angiography;
* Heart valve damage was confirmed by heart ultrasound, which is subject to surgical correction (aortic stenosis of III degree with a gradient on the aortic valve of more than 42 mmHg, aortic insufficiency III, mitral valve stenosis II-III, mitral regurgitation II-III)
* Patient consent to participate in the study;
* Women who have a negative pregnancy test and use effective contraception throughout the study and for 3 weeks after its completion, or women who are unable to have children (women who have undergone a hysterectomy (removal of the uterus) or tubal ligation, women with a clinical diagnosis of infertility) or are menopausal for more than 1 year (absence of menstruation for at least 12 months). Adequate methods of contraception include: surgical sterilization, double barrier method of contraception, local contraception;

Exclusion Criteria:

* Refusal to participate;
* Hypersensitivity to propofol, dexmedetomidine;
* Prolonged mechanical ventilation in case of surgical complications (bleeding, inadequate perfusion of the myocardium);
* Occurred ischemic stroke;
* History of the ischemic stroke;
* History of the neurodegenerative diseases;
* History of the mental disorders;
* Use of neuroleptics, antidepressants for the last 5 years;
* History of the cardiac surgery in the past;
* Patients with chronic pulmonary disease (GOLD 3-4)
* Patients with asthma (moderate or severe),
* Participation in any other clinical trial;
* Gastric or duodenal ulcer with risk of bleeding;
* Chronic renal failure (ClCr less than 50 ml / h)
* Acute renal failure that occurred during surgery (ClCr less than 50 ml / h, or a decrease in the rate of diuresis to 0.1 ml / h in the first 4 hours after surgery and does not respond to diuretic therapy)
* Chronic hepatic insufficiency if there are laboratory signs of hypo coagulation without the use of anticoagulant therapy (INR> 1.5)
* If the patient has not stopped taking anticoagulants or antiplatelet agents in the preoperative period: warfarin 5 days before surgery, clopidogrel 5-7 days before surgery, xarelto / pradaxa 3 days before surgery),
* History of the hematological disease;
* Alcohol abuse in the anamnesis (3-4 times a week).
* Condition after chemotherapy; Pregnancy, lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
hospital LOS | from admission to discharge ( up to 20 days)
  measure at days
ICU LOS | before discharging from ICU to the ward ( up to 7 days)
  measure at days

SECONDARY OUTCOMES:
difference in ICU LOS in patients with vasopressors and without vasopressors | before discharging from ICU to the ward ( up to 7 days
  measure at days

OTHER OUTCOMES:
difference in hospital LOS in patients with vasopressors and without vasopressors | from admission to discharge ( up to 20 days)
  measure at days

CONTACTS AND LOCATIONS:
Overall Officials: Yelyzaveta Plechysta, Principal Investigator — Chief of the anesthesia department
Locations (1):
- Medical Network Dobrobut, Kyiv, Ukraine